CLINICAL TRIAL: NCT01885884
Title: A Pilot Trial of an Embedded Collaborative Model of Supportive Care for Pancreatic Cancer
Brief Title: Supportive Care Intervention-Pancreas
Acronym: SCI-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Yael Schenker, MD, MAS, Assistant Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO13020507
Record Dates: First submitted 2013-06-07; First posted 2013-06-25 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Advanced Pancreatic Cancer
Keywords: Supportive Care; Palliative Care; Pancreatic Cancer; Embedded, coordinated model of supportive care within oncology care; Patient and Caregiver support
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supportive Care Intervention (Experimental): Monthly (minimum) patient & caregiver visits with a Supportive Care physician, embedded within their standard oncological care (through collaboration with oncology providers).
  Interventions: Behavioral: Embedded Supportive Care
- Usual Care (No Intervention): Participants will receive standard oncology care from their oncology providers.

INTERVENTIONS:
Behavioral: Embedded Supportive Care
  Arms: Supportive Care Intervention

SUMMARY:
This is a pilot, randomized controlled trial of an embedded collaborative model of supportive care designed to improve quality of life and decrease use of unwanted healthcare services at the end of life for patients with advanced pancreatic cancer. We will enroll 30 patients who are receiving treatment at the Hillman Cancer Center for recently diagnosed, locally advanced or metastatic pancreatic adenocarcinoma, as well as their accompanying caregivers and providers. Patients will be randomized to receive either the supportive care intervention or usual care. The purpose of this study is to refine an embedded collaborative model of supportive care and to develop protocols for recruitment, randomization, and longitudinal data collection.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  * Adults (≥ 18 years old)
  * Pathologically-confirmed locally advanced or metastatic pancreatic adenocarcinoma diagnosed within the past 8 weeks
  * Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 (asymptomatic), 1 (symptomatic but fully ambulatory), or 2 (symptomatic and in bed <50% of the day)
  * Planning to receive continued care from an oncologist at the Hillman Cancer Center
  * Accompanied by a caregiver (family member or friend) at the first visit
* Caregivers:

  * Adults (>= 18 years old)
  * Family member or friend of an eligible patient

Exclusion Criteria:

* Patients:

  * Unable to read and respond to questions in English
  * Not planning to receive continued care from an oncologist at the Hillman Cancer Center
  * Pancreatic neuroendocrine cancer
* Caregivers:

  * Unable to read and respond to questions in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
trial feasibility | up to 2 years
  We will assess trial feasibility by monitoring number of eligible patients per clinic day, contact rates, interest rates, enrollment rates, randomization rates, intervention visit completion rates, and outcome assessment completion rates.
acceptability of intervention participation | 3 months (+/- 3 weeks) from patient enrollment
  We will report the percentage of patients and caregivers who found the intervention acceptable.
intervention fidelity | Up to 2 years
  We will use post-visit checklists to characterize the number and types of recommended topics covered during each supportive care intervention visit.
perceived effectiveness | 3 months (+/- 3 weeks) from patient enrollment
  We will report the percentage of patients and caregivers who perceived the intervention to be effective for treating symptoms, understanding their illness, coping, and planning for the future.

SECONDARY OUTCOMES:
change in patient quality of life | baseline (enrollment) to 3 months (+/- 3 weeks) after enrollment
  We will summarize range and distribution of change in patient quality of life from baseline to 3 months using the Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep). Because this is a pilot trial, we will not conduct formal tests of efficacy.
patient healthcare utilization | up to 2 years
  We will summarize range and distribution of the following patient healthcare utilization outcomes: number and types of chemotherapy regimens, frequency and timing of chemotherapy regimens, number and length (days) of hospital admissions, number and length (days) of ICU admissions, number of emergency department visits, frequency and timing (days before death) of hospice use, place of death. Because this is a pilot trial, we will not conduct formal tests of efficacy.
patient quality of life | 3 months (+/- 3 weeks) from patient enrollment
  We will summarize range and distribution of patient quality of life at 3 months using the FACT-Hep scale. Because this is a pilot trial, we will not conduct formal tests of efficacy.

OTHER OUTCOMES:
patient illness understanding and care preferences | 3 months (+/- 3 weeks) from patient enrollment
  We will assess range and distribution of patient illness understanding using validated questions about patients' perceptions of curability, life expectancy, acknowledgement of whether or not s/he has a terminal illness, and preferences for comfort-oriented vs life-prolonging treatment. Because this is a pilot trial, we will not conduct formal tests of efficacy.
change in patient anxiety symptoms | baseline (enrollment) to 3 months (+/- 3 weeks) after enrollment
  We will assess change in patient anxiety symptoms with the Hospital Anxiety and Depression Scale (HADS) administered at baseline and 3 months. HADS scores will be compiled to assess range and distribution. Because this is a pilot trial, we will not conduct formal tests of efficacy.
change in patient distress | baseline (time of enrollment) to 3 months (+/- 3 weeks) after enrollment
  We will summarize range and distribution of change in patient distress responses from baseline to 3 months, collected with the National Comprehensive Cancer Network (NCCN) Distress Thermometer tool, where patients rate their distress on a visual guide from 0, 'no distress' to 10, 'extreme distress.' Scores will be compiled to assess range and distribution at 3-months. Because this is a pilot trial, we will not conduct formal tests of efficacy.
change in patient depressive symptoms | baseline (enrollment) to 3 months (+/- 3 weeks) after enrollment
  We will assess change in patient depression from baseline to 3 months with the Hospital Anxiety and Depression Scale (HADS) and the Primary Care Evaluation of Mental Disorders: Patient Health Questionnaire (PRIME-MD PHQ-9). HADS and PHQ-9 depression scores will be compiled to assess range and distribution at baseline and 3 months. Because this is a pilot trial, we will not conduct formal tests of efficacy.
change in caregiver distress | baseline (enrollment) to 3 months (+/- 3 weeks) after enrollment
  We will summarize range and distribution of change in caregiver distress responses from baseline to 3 months, collected with the National Comprehensive Cancer Network (NCCN) Distress Thermometer tool. Because this is a pilot trial, we will not conduct formal tests of efficacy.
change in caregiver burden | baseline (enrollment) to 3 months (+/- 3 weeks) after enrollment
  We will summarize the range and distribution of the reported change in caregiving burden from baseline to 3 months, collected with the Zarit Burden Interview and Family Member Concerns scale. Because this is a pilot trial, we will not conduct formal tests of efficacy.
caregiver grief | 1-3 months after death of enrolled patient
  We will assess caregiver grief after the death of their loved one (enrolled patient), if the patient dies during study participation and up to 2-year follow up. We will use the Inventory of Complicated Grief to assess how much and how often caregivers are affected by the loss of their loved one and summarize the range and distribution of this data. Because this is a pilot study, we will not conduct formal tests of efficacy.
change in caregiver anxiety symptoms | baseline (enrollment) to 3 months (+/- 3 weeks) after enrollment
  We will assess change in caregiver anxiety symptoms from baseline to 3 months with the Hospital Anxiety and Depression Scale (HADS). HADS scores will be compiled to assess range and distribution. Because this is a pilot trial, we will not conduct formal tests of efficacy.
change in caregiver depressive symptoms | baseline (enrollment) to 3 months (+/- 3 weeks) after enrollment
  We will assess change in caregiver depressive symptoms from baseline to 3 months with the Hospital Anxiety and Depression Scale (HADS). HADS scores will be compiled to assess range and distribution. Because this is a pilot trial, we will not conduct formal tests of efficacy.
caregiver perceptions of circumstances surrounding death and preparedness for death | 1-3 months after death of enrolled patient
  We will assess caregiver perceptions of circumstances surrounding death and preparedness for death using four previously validated questions. We will summarize range and distribution of responses. Because this is a pilot trial, we will not conduct formal tests of efficacy.
quality of life of seriously ill patients | 3 months (+/- 3 weeks) after enrollment
  We will summarize range and distribution of patient quality of life using the Quality of Life - Seriously Ill Patients (QUAL-E) score. Because this is a pilot trial, we will not conduct formal tests of efficacy.
patient emotional acceptance of illness | 3 months (+/- 3 weeks) after enrollment
  We will summarize range and distribution of patient emotional acceptance of illness using the PEACE Scale. Because this is a pilot trial, we will not conduct formal tests of efficacy.
patient anxiety | 3 months (+/- 3 weeks) after enrollment
  We will summarize range and distribution of patient anxiety using the Hospital Anxiety and Depression Scale (HADS). Because this is a pilot trial, we will not conduct formal tests of efficacy.
patient distress | 3 months (+/- 3 weeks) after enrollment
  We will summarize range and distribution in patient distress responses, collected with the National Comprehensive Cancer Network (NCCN) Distress Thermometer tool, where patients rate their distress on a visual guide from 0, 'no distress' to 10, 'extreme distress.' Because this is a pilot trial, we will not conduct formal tests of efficacy.
patient depression | 3 months (+/- 3 weeks) after enrollment
  We will assess patient depression from with the Hospital Anxiety and Depression Scale (HADS) and the Primary Care Evaluation of Mental Disorders: Patient Health Questionnaire (PRIME-MD PHQ-9). HADS and PHQ-9 depression scores will be compiled to assess range and distribution. Because this is a pilot trial, we will not conduct formal tests of efficacy.
caregiver distress | 3 months (+/- 3 weeks) after enrollment
  We will summarize range and distribution in caregiver distress responses, collected with the National Comprehensive Cancer Network (NCCN) Distress Thermometer tool. Because this is a pilot trial, we will not conduct formal tests of efficacy.
caregiver burden | 3 months (+/- 3 weeks) after enrollment
  We will summarize the range and distribution of the reported caregiving burden, collected with the Zarit Burden Interview and Family Member Concerns scale. Because this is a pilot trial, we will not conduct formal tests of efficacy.
caregiver anxiety symptoms | 3 months (+/- 3 weeks) after enrollment
  We will assess caregiver anxiety symptoms with the Hospital Anxiety and Depression Scale (HADS). HADS scores will be compiled to assess range and distribution. Because this is a pilot trial, we will not conduct formal tests of efficacy.
caregiver depressive symptoms | 3 months (+/- 3 weeks) after enrollment
  We will assess caregiver depressive symptoms with the Hospital Anxiety and Depression Scale (HADS). HADS scores will be compiled to assess range and distribution. Because this is a pilot trial, we will not conduct formal tests of efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Yael Schenker, MD, MAS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute (UPCI), Hillman Cancer Center, Pittsburgh, Pennsylvania, United States